CLINICAL TRIAL: NCT06098872
Title: Pilot Study on the Efficacy of MEK1/MEK2 Inhibitor Trametinib in Patients With Surgical Unruptured Arteriovenous Malformations
Brief Title: Pilot Study on Trametinib for Surgical Unruptured AVMs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5463; OZUHN-017 (Other: Ozmosis)
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-10

CONDITIONS: Arteriovenous Malformations
Keywords: Trametinib; Mitogen-activated-protein-kinase (MEK) inhibitor
MeSH Terms: conditions — Arteriovenous Malformations | interventions — trametinib

STUDY DESIGN:
Intervention Model Description: This is an open-label pilot study assessing the potential efficacy of Trametinib in improving AVM angioarchitecture for patients who are already planned to undergo surgical resection as part of their standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Oral Trametinib (Experimental): Participants will receive oral Trametinib once daily for up to 60 days prior to their elective surgery
  Interventions: Drug: Trametinib tablet

INTERVENTIONS:
Drug: Trametinib tablet — Drug is supplied in 2mg and 0.5 mg tablets

SUMMARY:
Arteriovenous malformation (AVM) is a tangle of abnormal vessels that can progress through life and cause significant bleeding, deformity, pain, and deficits in day-to-day activities. Surgery is a common treatment option for patients with AVMs where the goal is to safely remove the entire AVM without causing complications. While any surgery has its potential risks, most of the potential modifiable risk factors relate to the AVM's structure, such as the AVM size or presence of high risk structural features seen on scans. The purpose of this pilot study is to see whether taking an oral medication called Trametinib can improve upon the AVM structure in adult patients before their scheduled surgery.

DETAILED DESCRIPTION:
The goal of this pilot clinical trial is to see whether an oral medication called Trametinib can be given to patients with arteriovenous malformations (AVMs) of the brain and body before surgery in order to make the AVM structure less risky for surgery.

The main questions it aims to answer are:

1. does taking Trametinib make the structure of the AVM less risky for surgery? This will determined by comparing the size and structure of the AVM on repeat scans before and after taking the drug.
2. does taking Trametinib reduce the blood flow to the AVM? This will be determined by quantifying the blood flow to the AVM with quantitative magnetic resonance imaging software.
3. is the drug well tolerated in this patient population? This will be determined by following for any side effects of the medication
4. how does the drug do what it is supposed to do clinically by looking at its effect at the cell level? This will be determined by taking a piece of the AVM that is removed at the time of surgery and running experiments in the lab to compare its structure and behaviour to other AVMs that were not treated with this medication.

Participants will first undergo screening tests to ensure they are candidates for the medication. They will take oral Trametinib once daily for a total of 60 days prior to their planned surgery. They will be monitored for side effects at days 15, 30 and 60. They will undergo routine scans prior to starting the drug and then again within 5 days of their last dose to see any changes made to the AVM structure after taking the drug. Lastly, at the time of surgery, a part of the AVM removed will be sent to our research lab to see what the drug is doing at the cell level to result in the changes we can see on the scans.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Confirmed diagnosis of an unruptured AVM Spetzler-Martin Lawton Young Grade equal to or less than 6 on magnetic resonance imaging (MRI), CT-angiogram (CTA) or angiogram, and clinical exam by a physician who is familiar with this condition at any time in patient's medical history.
3. Planned surgical resection of AVM at University Health Network within the acceptable window defined by the study calendar (i.e. after the indicated study drug dosing period and approximate week-long follow up).
4. Patients must not have received an investigational drug within the 4 weeks prior to study enrolment.
5. Patients who have previously received biologic therapy treatment must have completed therapy at least 14 days prior to study enrolment.
6. Patients who have previously received myelosuppressive chemotherapy must have completed therapy at least 28 days prior to study enrolment.
7. Patients on anticoagulants must have stopped treatment within 7 days of starting Trametinib.
8. Patient is able to swallow oral medication and/or retain oral medication via G tube.
9. Patients of childbearing potential (as assessed by their local Investigator) and fertile men who are sexually active must agree to the use of 2 forms of contraception (as discussed with the overseeing physician) throughout the period of study treatment and for 16 weeks after last dose of study drug. They are not allowed to donate ova or sperm for up to 16 weeks after the last dose of study drug.

Exclusion Criteria:

1. AVM due to known germline mutation such as phosphatase and tensin homolog (PTEN) or known history of familial AVM syndromes.
2. Received prior map kinase (MEK) inhibitor therapy.
3. Known allergy or contraindication to MEK inhibitor treatment.
4. Patients who have undergone major surgery, as defined by the overseeing Investigator, within 28 days prior to study enrolment or who have not recovered from side effects of such a procedure.
5. Patients that are currently pregnant or breastfeeding.
6. A known history of coagulopathy and/or current use of anticoagulant therapy.
7. International normalized ratio (INR) > 1.5 within 7 days of enrolment.
8. Left ventricular ejection fraction (LVEF) <50%, or any ECG abnormalities within 7 days of enrolment.
9. Retinal vein occlusion, serous retinopathy or glaucoma diagnosed within 1 month of enrolment.
10. Diagnosis of significant liver failure (Child-Pugh score 2+) within 7 days of enrolment.
11. Rhabdomyolysis (creatinine kinase (CK) >5x ULN) within 7 days of enrolment.
12. Patients with known risk factors for gastrointestinal perforation (prior perforation, diverticulitis, metastases to the gastrointestinal tract and concomitant use of medications with a recognized risk of gastrointestinal perforation
13. Positive covid-19 polymerase chain reaction (PCR) test within 7 days of enrolment.
14. Patient is unwilling or unable to comply with study requirements.
15. Unstable health status that may interfere with completing the study, as assessed by the overseeing Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Radiological response by independent central review at day 60 or 5 days after last dose, whichever comes first | screening, Day 60 or 5 days after last dose (whichever comes first)
  as defined by one or more of the following: (1) at least 20% reduction in the volume of the AVM confirmed on repeat imaging, (2) resolution of angiographic weak points, or (3) resolution of AVM induced parenchymal changes by independent central review.

SECONDARY OUTCOMES:
Safety of Trametinib in surgical AVM population | screening, Day 15, 30, 60, within 1 week of surgery and up to 30 days after final dose
  Participants will be followed serially for the presence of adverse events, including their type, severity, and need for dose modifications or interruptions
Change from baseline in symptomatology and functional performance | screening, day 15, 30, and 60
  Participants will be followed serially for any changes in self-reported clinical symptoms or signs, and for any changes in functional outcome with the modified Rankin Scale (mRS) (scale from 0 to 6, with increasing score representing worse functional status)
Change from baseline in AVM blood flow | screening, day 60 or 5 days after final dose (whichever comes first)
  The blood flow to the AVM will be objectively compared over time after Trametinib dosing with serial quantitative magnetic resonance angiography imaging
Effect of Trametinib on AVM pathobiology | time of surgery
  The documentation of signaling pathways identified in AVM tissues after Trametinib drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Radovanovic, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansur A, Radovanovic I. Vascular malformations: An overview of their molecular pathways, detection of mutational profiles and subsequent targets for drug therapy. Front Neurol. 2023 Feb 10;14:1099328. doi: 10.3389/fneur.2023.1099328. eCollection 2023. PMID 36846125
- [Background] Nikolaev SI, Fish JE, Radovanovic I. Somatic Activating KRAS Mutations in Arteriovenous Malformations of the Brain. N Engl J Med. 2018 Apr 19;378(16):1561-1562. doi: 10.1056/NEJMc1802190. No abstract available. PMID 29669234
- [Background] Fish JE, Flores Suarez CP, Boudreau E, Herman AM, Gutierrez MC, Gustafson D, DiStefano PV, Cui M, Chen Z, De Ruiz KB, Schexnayder TS, Ward CS, Radovanovic I, Wythe JD. Somatic Gain of KRAS Function in the Endothelium Is Sufficient to Cause Vascular Malformations That Require MEK but Not PI3K Signaling. Circ Res. 2020 Aug 28;127(6):727-743. doi: 10.1161/CIRCRESAHA.119.316500. Epub 2020 Jun 17. PMID 32552404
- [Background] Hong T, Yan Y, Li J, Radovanovic I, Ma X, Shao YW, Yu J, Ma Y, Zhang P, Ling F, Huang S, Zhang H, Wang Y. High prevalence of KRAS/BRAF somatic mutations in brain and spinal cord arteriovenous malformations. Brain. 2019 Jan 1;142(1):23-34. doi: 10.1093/brain/awy307. PMID 30544177
- [Background] Nicholson CL, Flanagan S, Murati M, Boull C, McGough E, Ameduri R, Weigel B, Maguiness S. Successful management of an arteriovenous malformation with trametinib in a patient with capillary-malformation arteriovenous malformation syndrome and cardiac compromise. Pediatr Dermatol. 2022 Mar;39(2):316-319. doi: 10.1111/pde.14912. Epub 2022 Jan 10. PMID 35014097
- [Background] Lekwuttikarn R, Lim YH, Admani S, Choate KA, Teng JMC. Genotype-Guided Medical Treatment of an Arteriovenous Malformation in a Child. JAMA Dermatol. 2019 Feb 1;155(2):256-257. doi: 10.1001/jamadermatol.2018.4653. PMID 30566190
- [Background] Edwards EA, Phelps AS, Cooke D, Frieden IJ, Zapala MA, Fullerton HJ, Shimano KA. Monitoring Arteriovenous Malformation Response to Genotype-Targeted Therapy. Pediatrics. 2020 Sep;146(3):e20193206. doi: 10.1542/peds.2019-3206. PMID 32859736
- [Background] Wright CJ, McCormack PL. Trametinib: first global approval. Drugs. 2013 Jul;73(11):1245-54. doi: 10.1007/s40265-013-0096-1. PMID 23846731
- [Background] Couto JA, Huang AY, Konczyk DJ, Goss JA, Fishman SJ, Mulliken JB, Warman ML, Greene AK. Somatic MAP2K1 Mutations Are Associated with Extracranial Arteriovenous Malformation. Am J Hum Genet. 2017 Mar 2;100(3):546-554. doi: 10.1016/j.ajhg.2017.01.018. Epub 2017 Feb 9. PMID 28190454